CLINICAL TRIAL: NCT06075862
Title: Postural Imbalance Amongst Elderly Patients With Symptomatic Lumbar Spinal Stenosis Before and After Decompressive Surgery
Brief Title: Balance Amongst Patients With Lumbar Spinal Stenosis
Acronym: B-ATLAS
Status: Recruiting | Type: Observational
Sponsor: Region Zealand (Other)
Collaborators: Region Syddanmark (Other)
Responsible Party: Principal Investigator, Oliver Bremerskov Zielinski, Principal Investigator, Region Zealand
Other Study IDs: B-ATLAS1; 010-0194/22-3000 (Registry Identifier: B-ATLAS)
Record Dates: First submitted 2023-09-11; First posted 2023-10-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Spinal stenosis; Elderly; Balance; Surgery
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with lumbar spinal stenosis: Patients diagnosed with lumbar spinal stenosis and referred to operation. Balance will be measured once in this group before operation, and four times again after operation.
  Interventions: Procedure: Decompressive surgery

INTERVENTIONS:
Procedure: Decompressive surgery — Decompressive lumbar spinal surgery

SUMMARY:
Lumbar spinal stenosis (LSS) is one of the most common degenerative diseases of the spinal column, with symptoms including low back pain which worsens with ambulation, poor balance, decreased activity due to pain, and a marked decrease in quality of life (QoL). Prevalence rises with age, and current treatment options range from varied conservative management strategies, to surgical intervention with decompression of neural structures.

While the effects of surgical decompression on back pain and QoL has been widely researched, the effects of surgery on patient balance is less well understood. Though patients generally have subjective improvements in this parameter after surgery, objective measurements in this patient group have been lacking.

This study aims to investigate the effects of decompressive surgery on postural balance in elderly patients with LSS. Measurements of postural balance will be taken before and after decompressive surgery, as well as with regular intervals during a two-year follow-up period.

A better understanding of the effect that LSS has on balance may lead to more patients being able to receive surgical treatment, which is hypothesized to lead to an increase in QoL and less perceived disability amongst this patient group.

DETAILED DESCRIPTION:
Disease Background:

While lumbar spinal stenosis (LSS) is one of the most common degenerative diseases of the spinal column, there is no universally accepted definition of LSS, and no accepted radiologic diagnostic criteria. LSS most often refers to a narrowing in the central canal of the vertebrae, the lateral recess, or the neural foramen. Changes to these can occur due to acquired degenerative spondylosis or spondylolisthesis, or more rarely due to conditions such as ankylosing spondylitis and space-occupying lesions, or congenital abnormalities. LSS can be classified according to anatomical location, etiology or severity of narrowing, though no validated classification has been published.

The lack of concrete definition has caused difficulties in estimating the prevalence of LSS. Studies using community-based sampling has shown a prevalence of acquired LSS, defined as a narrowing of the central canal to ≤ 10mm in the anterior-posterior direction, of 7.3%. The prevalence has been shown to rise with age, from 4.0% affected at < 40 years of age, to 14.3% amongst patients ≥ 60. No significant differences have been observed in overall prevalence according to gender, although there seems to be a slightly higher prevalence amongst elderly females than males.

Although LSS is often asymptomatic, common symptoms of LSS include low back pain, which worsens with prolonged ambulation, lumbar extension and standing, and which is relieved by rest and forward flexion, as well as lumbar radiculopathy. Patients may also complain of poor balance, and physical examination findings may include a wide-based gait and abnormal Romberg results. Symptoms are thought to occur due to compression of microvascular structures in the nerves, allowing for neural ischemia and defects in nerve conduction, and venous pooling resulting in inadequate oxygenation and metabolite accumulation.

Current treatment options for LSS range across both conservative and surgical management strategies. Conservative management has traditionally been regarded as first-line treatment, with a combination approach of physical therapy and pharmacological treatment with NSAIDs and analgesics. Epidural steroid injections have been used for symptom management, though with limited short and long-term benefits. Surgical management is often indicated in patients with ongoing pain despite attempts at conservative management for 3-6 months. Choice of surgical strategy to relieve the pressure on the neural structures depends on the anatomical location of stenosis and number of stenotic segments, as well as the intraoperative assessment of stability.

The effect of surgical decompression on disability, leg pain and back pain has been widely evaluated, but studies of the effect on postural control are sparse. The present study aims to investigate the effect of surgical decompression of symptomatic lumbar spinal stenosis on postural control by assessment of sway measures before and after surgery.

Postural Balance:

Mechanical balance is defined according to Newton's first law, stating that an object is at equilibrium (balanced) when the forces acting upon it are zero. When considering the balance of an object, the objects centre of gravity (COG) and its base of support (BOS) must be examined. For an object to remain balanced, a vertical line drawn from the COG to the objects BOS, the point of intersection defined as the centre of pressure (COP), must lie within the objects BOS. When the COP goes beyond the BOS, objects become unbalanced and may topple. If in a state of imbalance, humans and animals have physiological compensatory mechanisms to ensure that their COP returns to lie within their BOS. The act of keeping the COP within the BOS is what is intuitively know as human balance.

No central definition of postural balance exists, but a widely cited definition is 'the act of maintaining, achieving or restoring a state of balance during any posture or activity'. Postural balance has previously been considered a summation of postural reflexes alongside sensory feedback mechanisms, with a single neural circuit system integrating somatosensory, vestibular, and visual systems to maintain equilibrium. However, efforts have been made to move away from this viewpoint, and the act of postural balance is now seen as an independent motor skill, incorporating complex physiological mechanisms as well as high-level somatosensory information processing, influenced by individual body schema and personal cognitive elements. Maintaining postural balance is now seen as a summation of two simultaneous and overlapping systems; one to control posture through tonic muscle activity, and one to maintain equilibrium when exposed to internal and external perturbations. Balance is hereby maintained using skeletal muscle with both phasic and tonic activity, with signals originating from distinct neural circuits including from the brain stem, cerebellum, motor cortex etc.

As of writing, no gold standard exists to measure balance, which has allowed a wide variety of techniques to be developed to measure postural balance skills amongst patients, and variables associated with postural control, either through instrumented or non-instrumented tests. Regarding the latter, expert consensus points to the use of the Berg Balance Scale or the Mini Balance Evaluation Systems Test when measuring postural balance in adult populations. However, while non-instrumented tests can give a gross indicator of postural balance, there exists a need for more granular analysis, which can be achieved using instrumented tests. The force platform remains the most widely used device for this purpose, allowing for the quantification of positional and dynamic variables associated with COP position, displacement, and trajectory.

The causes of imbalance are many. Any deficit or pathology relating to somatosensory, motor control or cognitive systems associated with postural control can lead to postural imbalance, including a wide range of pathological conditions such as visuo-vestibular and neurodegenerative diseases, as well as orthopaedic and rheumatological diseases of the musculoskeletal system. While aging itself does not seem to be an independent risk factor for postural imbalance, age-related changes in physiology have been linked to degeneration in postural imbalance, including decreased visual acuity, somatosensory loss, vestibular dysfunction, lower extremity muscle weakness and cognitive impairment.

As mentioned, objects which become unbalanced due to COP dislocation beyond the objects BOS may fall. Balance impairment, measured by dynamic variables using force plates as well as non-instrumental tests, have been shown to be predictors of falls amongst elderly. Falls represent a large healthcare burden, having serious risk of related injury, rising prevalence with age and being a significant cause of mortality amongst elderly. Furthermore, falls have been shown to be an independent risk factor of functional decline. As such, fall prevention is a topic of both national and international interest.

Spinal stenosis has shown to be a risk factor for both postural imbalance as well as a risk factor for falls. Previous studies have made efforts to quantify the effects of decompressive surgery on postural imbalance, though have remained limited by number of patients and short follow-up regimes, as well as lacking correlation between measurements of postural imbalance and risk of falls.

Wii Balance Board:

The Wii Balance Board (WBB), first released in 2007, has gained popularity as a low-cost, portable force-plate transducer, to use in postural balance assessment. It contains four transducers used to measure COP, as well as a scale to measure weight, and was originally used as a video game controller for the game WiiFit. Although capable of providing an intrinsic WiiFit Stillness score, this has shown limited usability in previous studies. However, using custom software, the WBB has been extensively validated against 'gold standard' laboratory-grade force plates, and shown to have good within-device and between-device reliability, as well as being a valid tool to measure balance amongst older adults. Work has been done to ensure that the WBB can be calibrated to minimize measurement error, and open-source algorithms exist for the calculation of positional and dynamic variables recorded by the WBB. While not recommended for clinical diagnostic measurements, the use of the WBB in longitudinal monitoring for research purposes remains viable.

Rationale of the study:

This study will be the first to correlate the effects of decompressive surgery in patients with symptomatic LSS with postural balance, and associated quality of life increases. Previous studies have been hampered by low power due to sampling size limitations, and short follow-up regimes, both of which is sought to be managed through multi-centre collaboration and inclusion, and a follow-up regime spanning two years from the time of surgery.

It is expected that the results of this study can facilitate an increased understanding of the role of postural balance when considering surgical management of symptomatic LSS patients, as well as enable targeted treatment of patients with postural imbalance and LSS.

Research question:

Do elderly patients with symptomatic LSS, who have undergone decompressive surgery, show an improvement in postural balance compared to pre-operative values?

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Referred to decompressive spinal surgery due to symptomatic lumbar spinal stenosis at ≥ 1 level
* Central canal LSS grade B or C (Schizas classification) at ≥ 1 level by Magnetic Resonance Imaging
* Minimum of 3 months of unsuccessful non-operative treatment

Exclusion Criteria:

* Signs of malignancy or infection in the spinal column
* Severe comorbidities incl. neurodegenerative conditions which may contribute to balance problems
* Revision surgery (previous decompression surgery at the same vertebral level)
* Spinal surgery up to 1 year prior to the date of inclusion
* Mini Mental State Exam (MMSE) score of ≤ 27 points
* Degenerative spondylolisthesis more than 3mm on pre-operative imaging diagnostics

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 65 years of age referred to decompressive surgery for lumbar spinal stenosis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Postural balance | Before surgery and 3, 6, 12 and 24 months after surgery
  Postural balance, measured by sway area of center of pressure (mm^2)

SECONDARY OUTCOMES:
Postural balance | Before surgery and 3, 6, 12 and 24 months after surgery
  Postural balance measured by mean center of pressure velocity in the anterior-posterior and medio-lateral plane (mm^2/s)
Quality of life | Before surgery and 3, 6, 12 and 24 months after surgery
  Subjective QoL, measured by European Quality of Life - 5 Dimensions score (EQ-5D) The EQ-5D consists of six questions regarding current perceived health status and quality of life.
  Questions 1 - 5 have a range of 1 to 3, lower is better. The answer to questions 6 is given on a scale of 0 to 100, where lower is better.
Functional disability | Before surgery and 3, 6, 12 and 24 months after surgery
  Subjective functional disability, measured by Zurich Claudication Questionnaire score (ZCQ) The ZCQ consists of 12 questions for all patients, and a further six questions for patients who have received treatment.
  The questionnaire is divided into three subscales:
  Symptom severity scale (questions 1 - 7): range of the score is 1 to 5, lower is better.
  Physical function scale (questions 8 - 12): range of the score is 1 to 4, lower is better.
  Satisfaction with treatment scale (questions 13 - 18): range of the score is 1 to 4, lower is better.
Quality of life | Before surgery and 3, 6, 12 and 24 months after surgery
  Subjective Quality-of-life, measured by the Short Form Health Survey (SF-36). The SF-36 is a short form questionnaire concerning patients perceived health and quality-of-life (QoL). It consists of 36 questions regarding various aspects of the patients health status, including current and past perceived physical and mental health, and subjective physical function.
  Questions 1,2 and 20 - 22 each have a range of 1 to 5, lower is better. Question 32 likewise has a range of 1 - 5, though where higher is better. Questions 3 - 12 have a range of 1 - 3, higher is better. Questions 13 - 19 have a range of 1 - 2, higher is better. Questions 23 - 31 and 33 - 36 have a range of 1 - 5. The better score depends on the specific question.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver B Zielinski, MD, Principal Investigator — Region Zealand
Locations (2):
- Denmark (2):
  - Ortopædkirurgisk afdeling, Sjællands Universitetshospital Køge, Køge
  - Rygcenter Syddanmark, Middelfart Sygehus, Middelfart

IPD SHARING:
Plan to Share IPD: Yes
All deidentified individual participant data collected during the trial will be made available to researchers who provide a methodologically sound proposal for use, subject to approval by the study authors.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: A deidentified copy of all individual participant data will be kept by the authors of the study for 10 years following study end. After this time period, the full data set will be archived by the Danish National Archives with no planned end date.
Access Criteria: Reasonable request for access can be made by writing to ozi@regionsjaelland.dk or rudb@regionsjaelland.dk in a time period consisting of 10 years after study end. After this period, requests for access can be made to the Danish National Archives at data@sa.dk.

REFERENCES:
- [Background] Binder DK, Schmidt MH, Weinstein PR. Lumbar spinal stenosis. Semin Neurol. 2002 Jun;22(2):157-66. doi: 10.1055/s-2002-36539. PMID 12524561
- [Background] Schroeder GD, Kurd MF, Vaccaro AR. Lumbar Spinal Stenosis: How Is It Classified? J Am Acad Orthop Surg. 2016 Dec;24(12):843-852. doi: 10.5435/JAAOS-D-15-00034. PMID 27849674
- [Background] Kalichman L, Cole R, Kim DH, Li L, Suri P, Guermazi A, Hunter DJ. Spinal stenosis prevalence and association with symptoms: the Framingham Study. Spine J. 2009 Jul;9(7):545-50. doi: 10.1016/j.spinee.2009.03.005. Epub 2009 Apr 23. PMID 19398386
- [Background] Yabuki S, Fukumori N, Takegami M, Onishi Y, Otani K, Sekiguchi M, Wakita T, Kikuchi S, Fukuhara S, Konno S. Prevalence of lumbar spinal stenosis, using the diagnostic support tool, and correlated factors in Japan: a population-based study. J Orthop Sci. 2013 Nov;18(6):893-900. doi: 10.1007/s00776-013-0455-5. Epub 2013 Aug 21. PMID 23963588
- [Background] Katz JN, Dalgas M, Stucki G, Katz NP, Bayley J, Fossel AH, Chang LC, Lipson SJ. Degenerative lumbar spinal stenosis. Diagnostic value of the history and physical examination. Arthritis Rheum. 1995 Sep;38(9):1236-41. doi: 10.1002/art.1780380910. PMID 7575718
- [Background] Lurie J, Tomkins-Lane C. Management of lumbar spinal stenosis. BMJ. 2016 Jan 4;352:h6234. doi: 10.1136/bmj.h6234. PMID 26727925
- [Background] Lee BH, Moon SH, Suk KS, Kim HS, Yang JH, Lee HM. Lumbar Spinal Stenosis: Pathophysiology and Treatment Principle: A Narrative Review. Asian Spine J. 2020 Oct;14(5):682-693. doi: 10.31616/asj.2020.0472. Epub 2020 Oct 14. PMID 33108834
- [Background] Mazanec DJ, Podichetty VK, Hsia A. Lumbar canal stenosis: start with nonsurgical therapy. Cleve Clin J Med. 2002 Nov;69(11):909-17. doi: 10.3949/ccjm.69.11.909. PMID 12430977
- [Background] Liu K, Liu P, Liu R, Wu X, Cai M. Steroid for epidural injection in spinal stenosis: a systematic review and meta-analysis. Drug Des Devel Ther. 2015 Jan 30;9:707-16. doi: 10.2147/DDDT.S78070. eCollection 2015. PMID 25678775
- [Background] Kovacs FM, Urrutia G, Alarcon JD. Surgery versus conservative treatment for symptomatic lumbar spinal stenosis: a systematic review of randomized controlled trials. Spine (Phila Pa 1976). 2011 Sep 15;36(20):E1335-51. doi: 10.1097/BRS.0b013e31820c97b1. PMID 21311394
- [Background] Sengupta DK, Herkowitz HN. Lumbar spinal stenosis. Treatment strategies and indications for surgery. Orthop Clin North Am. 2003 Apr;34(2):281-95. doi: 10.1016/s0030-5898(02)00069-x. PMID 12914268
- [Background] Pollock AS, Durward BR, Rowe PJ, Paul JP. What is balance? Clin Rehabil. 2000 Aug;14(4):402-6. doi: 10.1191/0269215500cr342oa. PMID 10945424
- [Background] Ivanenko Y, Gurfinkel VS. Human Postural Control. Front Neurosci. 2018 Mar 20;12:171. doi: 10.3389/fnins.2018.00171. eCollection 2018. PMID 29615859
- [Background] Paillard T, Noe F. Techniques and Methods for Testing the Postural Function in Healthy and Pathological Subjects. Biomed Res Int. 2015;2015:891390. doi: 10.1155/2015/891390. Epub 2015 Nov 12. PMID 26640800
- [Background] Sibley KM, Howe T, Lamb SE, Lord SR, Maki BE, Rose DJ, Scott V, Stathokostas L, Straus SE, Jaglal SB. Recommendations for a core outcome set for measuring standing balance in adult populations: a consensus-based approach. PLoS One. 2015 Mar 13;10(3):e0120568. doi: 10.1371/journal.pone.0120568. eCollection 2015. PMID 25768435
- [Background] Quijoux F, Nicolai A, Chairi I, Bargiotas I, Ricard D, Yelnik A, Oudre L, Bertin-Hugault F, Vidal PP, Vayatis N, Buffat S, Audiffren J. A review of center of pressure (COP) variables to quantify standing balance in elderly people: Algorithms and open-access code. Physiol Rep. 2021 Nov;9(22):e15067. doi: 10.14814/phy2.15067. PMID 34826208
- [Background] Kim SD, Allen NE, Canning CG, Fung VS. Postural instability in patients with Parkinson's disease. Epidemiology, pathophysiology and management. CNS Drugs. 2013 Feb;27(2):97-112. doi: 10.1007/s40263-012-0012-3. PMID 23076544
- [Background] Ruhe A, Fejer R, Walker B. Center of pressure excursion as a measure of balance performance in patients with non-specific low back pain compared to healthy controls: a systematic review of the literature. Eur Spine J. 2011 Mar;20(3):358-68. doi: 10.1007/s00586-010-1543-2. Epub 2010 Aug 19. PMID 20721676
- [Background] Boucher P, Descarreaux M, Normand MC. Postural control in people with osteoarthritis of the cervical spine. J Manipulative Physiol Ther. 2008 Mar;31(3):184-90. doi: 10.1016/j.jmpt.2008.02.008. PMID 18394494
- [Background] Fujimoto C, Egami N, Kinoshita M, Sugasawa K, Yamasoba T, Iwasaki S. Postural stability in vestibular neuritis: age, disease duration, and residual vestibular function. Laryngoscope. 2014 Apr;124(4):974-9. doi: 10.1002/lary.24342. Epub 2013 Oct 5. PMID 23929712
- [Background] Alexander NB. Postural control in older adults. J Am Geriatr Soc. 1994 Jan;42(1):93-108. doi: 10.1111/j.1532-5415.1994.tb06081.x. No abstract available. PMID 8277123
- [Background] Quijoux F, Vienne-Jumeau A, Bertin-Hugault F, Zawieja P, Lefevre M, Vidal PP, Ricard D. Center of pressure displacement characteristics differentiate fall risk in older people: A systematic review with meta-analysis. Ageing Res Rev. 2020 Sep;62:101117. doi: 10.1016/j.arr.2020.101117. Epub 2020 Jun 19. PMID 32565327
- [Background] Muir SW, Berg K, Chesworth B, Speechley M. Use of the Berg Balance Scale for predicting multiple falls in community-dwelling elderly people: a prospective study. Phys Ther. 2008 Apr;88(4):449-59. doi: 10.2522/ptj.20070251. Epub 2008 Jan 24. PMID 18218822
- [Background] Tinetti ME, Williams CS. The effect of falls and fall injuries on functioning in community-dwelling older persons. J Gerontol A Biol Sci Med Sci. 1998 Mar;53(2):M112-9. doi: 10.1093/gerona/53a.2.m112. PMID 9520917
- [Background] Muir SW, Berg K, Chesworth B, Klar N, Speechley M. Quantifying the magnitude of risk for balance impairment on falls in community-dwelling older adults: a systematic review and meta-analysis. J Clin Epidemiol. 2010 Apr;63(4):389-406. doi: 10.1016/j.jclinepi.2009.06.010. Epub 2009 Sep 9. PMID 19744824
- [Background] Kim HJ, Chun HJ, Han CD, Moon SH, Kang KT, Kim HS, Park JO, Moon ES, Kim BR, Sohn JS, Shin SY, Jang JW, Lee KI, Lee HM. The risk assessment of a fall in patients with lumbar spinal stenosis. Spine (Phila Pa 1976). 2011 Apr 20;36(9):E588-92. doi: 10.1097/BRS.0b013e3181f92d8e. PMID 21242866
- [Background] Truszczynska A, Drzal-Grabiec J, Trzaskoma Z, Rapala K, Tarnowski A, Gorniak K. A comparative analysis of static balance between patients with lumbar spinal canal stenosis and asymptomatic participants. J Manipulative Physiol Ther. 2014 Nov-Dec;37(9):696-701. doi: 10.1016/j.jmpt.2014.09.003. Epub 2014 Sep 26. PMID 25267441
- [Background] Truszczynska A, Drzal-Grabiec J, Trzaskoma Z, Rachwal M, Rapala K, Gorniak K. Static balance after surgical decompression of lumbar spinal canal stenosis. J Back Musculoskelet Rehabil. 2015;28(4):865-71. doi: 10.3233/BMR-150646. PMID 26519120
- [Background] Kneis S, Bruetsch V, Dalin D, Hubbe U, Maurer C. Altered postural timing and abnormally low use of proprioception in lumbar spinal stenosis pre- and post- surgical decompression. BMC Musculoskelet Disord. 2019 May 1;20(1):183. doi: 10.1186/s12891-019-2497-0. PMID 31043162
- [Background] Iversen MD, Kale MK, Sullivan JT Jr. Pilot case control study of postural sway and balance performance in aging adults with degenerative lumbar spinal stenosis. J Geriatr Phys Ther. 2009;32(1):15-21. doi: 10.1519/00139143-200932010-00004. PMID 19856631
- [Background] Negus JJ, Cawthorne D, Clark R, Negus O, Xu J, March PL, Parker D. Validity and reliability of the Nintendo Wii Fit Stillness score for assessment of standing balance. Asia Pac J Sports Med Arthrosc Rehabil Technol. 2018 Sep 14;15:29-34. doi: 10.1016/j.asmart.2018.09.001. eCollection 2019 Jan. PMID 30581757
- [Background] Reed-Jones RJ, Dorgo S, Hitchings MK, Bader JO. WiiFit Plus balance test scores for the assessment of balance and mobility in older adults. Gait Posture. 2012 Jul;36(3):430-3. doi: 10.1016/j.gaitpost.2012.03.027. Epub 2012 Apr 23. PMID 22534562
- [Background] Clark RA, Bryant AL, Pua Y, McCrory P, Bennell K, Hunt M. Validity and reliability of the Nintendo Wii Balance Board for assessment of standing balance. Gait Posture. 2010 Mar;31(3):307-10. doi: 10.1016/j.gaitpost.2009.11.012. Epub 2009 Dec 11. PMID 20005112
- [Background] Scaglioni-Solano P, Aragon-Vargas LF. Validity and reliability of the Nintendo Wii Balance Board to assess standing balance and sensory integration in highly functional older adults. Int J Rehabil Res. 2014 Jun;37(2):138-43. doi: 10.1097/MRR.0000000000000046. PMID 24445863
- [Background] Leach JM, Mancini M, Peterka RJ, Hayes TL, Horak FB. Validating and calibrating the Nintendo Wii balance board to derive reliable center of pressure measures. Sensors (Basel). 2014 Sep 29;14(10):18244-67. doi: 10.3390/s141018244. PMID 25268919
- [Derived] Zielinski OB, Hallager DW, Jensen KY, Carreon L, Andersen MO, Diederichsen LP, Bech RD. Multicentre investigation on the effect of decompressive surgery on Balance and physical ActiviTy Levels amongst patients with lumbar Spinal stenosis (B-ATLAS): protocol for a prospective cohort study. BMJ Open. 2024 Sep 23;14(9):e085667. doi: 10.1136/bmjopen-2024-085667. PMID 39313282